CLINICAL TRIAL: NCT06498700
Title: Intraoperative Subanesthetic Ketamine Versus Dexmedetomidine Infusion for Prevention of Post-traumatic Stress Disorder After Traumatic Brain Surgeries: A Randomized Trial
Brief Title: Intraoperative Subanesthetic Ketamine Versus Dexmedetomidine Infusion for Prevention of Post-traumatic Stress Disorder After Traumatic Brain Surgeries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 440
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Subanesthetic Ketamine Dexmedetomidin
Keywords: Ketamine, Dexmedetomidine ,Post-traumatic Stress Disorder , traumatic Brain surgeries
MeSH Terms: interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine(K) (Experimental): 0.5 mg/kg/h ketamine infusion
  Interventions: Drug: ketamine
- dexmedetomidine(D) (Experimental): 0.1 ug/kg/h dexmedetomidine infusion
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: ketamine — 0.5 mg/kg/h ketamine infusion
  Arms: Ketamine(K)
Drug: dexmedetomidine — 0.1 ug/kg/h dexmedetomidine infusion
  Arms: dexmedetomidine(D)

SUMMARY:
Prevention of Post-traumatic Stress Disorder after traumatic Brain surgeries by using either subanesthetic ketamine or dexmedetomidine infusion.

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double blind manner into two equal groups (K group and D group). Using computer generated randomization table; each group consists of 26 patients: K group (n=26): Patient will receive with 0.5 mg/kg/h ketamine infusion. D group (n=26): Patient will receive 0.1 ug/kg/h dexmedetomidine infusion.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-60 years old.Body mass index of less than or equal 35.American Society of I and II.Duration of surgery not more than 3 hours.

Exclusion Criteria:

Known hypersensitivity to dexmedetomidine or ketamine. Hemorrhagic shock decompensation.History of alcohol or drug abuse.History of neurologic or psychiatric diseases Advanced renal ,liver or cardiovascular disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
(PTSD) | 6 months
  To measure the change in PTSD symptom severity using the PTSD Checklist

SECONDARY OUTCOMES:
VAS | (24 hours, 48 hours, and 1 month)
  postoperative pain
postoperative delirium | twice daily for 3 days
  using the confusion assessment method criteria

CONTACTS AND LOCATIONS:
Overall Officials: marwa M Medhat, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No